CLINICAL TRIAL: NCT01180959
Title: A Phase II Trial of Erlotinib Plus Bevacizumab in Advanced Hepatocellular Carcinoma as a Second-line Therapy in Patients Who Have Received First-line Sorafenib Therapy (AVF4572)
Brief Title: Erlotinib Plus Bevacizumab in Hepatocellular Carcinoma (HCC) as Second-line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0260; NCI-2011-00723 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Liver Cancer
Keywords: Advanced Liver Cancer; primary neoplasm of the liver; Erlotinib; Bevacizumab; Hepatocellular Carcinoma; HCC; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; OSI-774; Tarceva
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erlotinib + Bevacizumab (Experimental): Erlotinib 150 mg by mouth once a day. Bevacizumab 10 mg/kg by vein once every 2 weeks on days 1 and 15 of each cycle. The first dose of bevacizumab will be given over about 90 minutes.
  Interventions: Drug: Bevacizumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg by vein once every 2 weeks on days 1 and 15 of each cycle. The first dose of bevacizumab will be given over about 90 minutes
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Erlotinib — 150 mg by mouth once a day.
  Other Names: OSI-774; Tarceva

SUMMARY:
The goal of this clinical research study is to learn if the combination of AvastinTM (bevacizumab) and Tarceva (erlotinib hydrochloride) can help to control advanced liver cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to block the growth of blood vessels that supply nutrients necessary for tumor growth. This may prevent or slow down the growth of cancer cells.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing. There is a commercially available form of the drug (called Tarceva) that is expected to be very similar to the erlotinib being used for this study, but it is possible that there may be some differences between the 2 formulations.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive the study drugs during 28-day "study cycles."

You will receive bevacizumab by vein on Days 1 and 15 of each cycle. The first dose of bevacizumab will be given over about 90 minutes. If you do not have a reaction to the drug, such as fever and/or chills, the next dose will be given over about 60 minutes. If you still have no reaction after the second dose, each dose after that will be given over about 30 minutes. If you experience a reaction to the bevacizumab, you may be given Tylenol® (acetaminophen) by mouth and/or an antihistamine by vein over 30 minutes before each dose to help minimize the risk of further reactions.

You will take 1 erlotinib hydrochloride tablet by mouth every day. You should take erlotinib hydrochloride in the morning with a full glass of water (6-8oz) at least 1 hour before or 2 hours after any food, grapefruit juice, vitamins, iron supplements, or other non-prescription drugs.

Study Visits:

On Day 1 of Cycle 2 and beyond:

* Blood (about 3 tablespoons) will be drawn for routine blood tests and to check how well the blood clots.
* Urine will be collected for routine testing. A 24-hour urine sample may be collected if needed. If a 24-hour urine sample is needed, you will be provided with a special container to collect the sample.
* You will be asked questions about any side effects you may have had and about any drugs you may be currently taking or have taken since you last saw the study doctor.
* You will have a complete physical exam, including measurements of weight and vital signs.
* Your performance status will be recorded.

On Day 15 of Cycle 2 and beyond, your vital signs will be recorded.

At the end of Cycle 2, 4, and every 2 cycles after that (Cycles 6, 8, 10, and so on):

°You will have CT/MRI scans of the abdomen and pelvis and chest scan (if the doctor thinks they are needed) to check the status of the disease.

Additional tests may be done during the study if the study doctor thinks it is necessary.

Length of Treatment:

You will receive bevacizumab and erlotinib hydrochloride for as long as you are benefitting. There is no maximum number of cycles that you can receive. If you experience severe side effects, the treatment on this study may be delayed, stopped, or the study doctor may give you smaller doses of the study drugs. You will be taken off study if the disease gets worse, the side effects are too severe, or your doctor thinks that it is in your best interest to stop receiving treatment.

End-of-Treatment Visit:

After you stop receiving all of the study drugs, you will return for an end-of-treatment visit. At this visit, the following tests and procedures will be performed:

* Blood (about 3 tablespoons) and urine will be collected for routine tests and to learn how well the blood clots.
* You will be asked questions about any side effects you may have had and about any drugs you may be currently taking or have taken since you last saw the study doctor.
* You will have a complete physical exam, including measurements of weight and vital signs.
* Your performance status will be recorded.
* CT and/or MRI scans of the abdomen and pelvis will be performed to check the status of the disease.

Follow-Up:

After the end-of-treatment visit, the study doctor will continue to review your medical records every 3 months until the study analysis is complete. You will also be called every 3 months for as long as the study doctor thinks is needed. During these phone calls, you will be asked about how you are doing and if you are experiencing any health problems. The phone call should take about 15 minutes. During the follow-up period, if the study doctor thinks it is necessary, you may be asked to come in for a clinic visit.

This is an investigational study. Bevacizumab is FDA approved and commercially available for the treatment of metastatic colon and rectal cancer. Erlotinib hydrochloride is FDA approved and commercially available for the treatment of lung cancer. The use of this drug combination in patients with advanced liver cancer is investigational.

Up to 44 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological or cytologically documented HCC not amenable to curative resection (documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable) or clinical diagnosis by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic subjects is required. For subjects without cirrhosis, histological or cytological confirmation is mandatory.
2. Patients must have measurable disease as per the modified RECIST criteria. Measurable target lesions are defined at baseline as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) >/= 20 mm using conventional techniques (CT or MRI) or >/= 10 mm using spiral CT scan. Lesion must not be chosen from a previously irradiated field, unless there has been documented disease progression in that field after irradiation.
3. Patients who have progressed on, or were intolerant to, one prior systemic therapy with sorafenib, completed ≥ 14 days prior to treatment day 1. Previous treatments also allowed that do not count as systemic therapy include: surgical resection, transarterial embolization/chemoembolization (TAE/TACE), radiofrequency ablation (RFA), percutaneous ethanol injection (PEI), provided that the lesion(s) to be evaluated in this study are separate from the previously treated lesions(s).
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= 2.
5. Childs-Pugh liver function status of A or B (only 7 points allowed).
6. Organ function: Absolute peripheral granulocyte count of >/= 1500 mm^3, platelet count of >/= 40,000 mm^3, hemoglobin >/= 10 gm/dL. Total bilirubin </= 2.0 gm/dL; serum albumin >/= 2.5 gm/dL; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) up to 5 X the upper limit of institutional normal (AST - 46 and ALT - 56); and prothrombin time prolonged not more than 3 seconds greater than institutional normal, once attempts to correct a prolonged PT have been made.
7. (Continuation of # 6) Patients who require full dose anticoagulation, who are otherwise eligible for this trial, are allowed to have an appropriately prolonged International Normalized Ratio (INR).
8. Negative serum pregnancy test in women with childbearing potential (those who are not surgically sterilized or who are not amenorrheic for >/= 12 months), within one week prior to initiation of treatment.
9. Men and women of childbearing potential must agree to use effective means of contraception prior to study entry and for at least 180 days after the last dose of study treatment. They must agree to use two forms of birth control, for example, barrier methods (such as a diaphragm, cervical cap, contraceptive sponge, female condom, or male condom), and an intrauterine device (IUD).
10. Age >/= 18 years. The agents bevacizumab and erlotinib have not been studied in pediatric patients, thus the doses to be used in this study cannot be assumed to be safe in children.
11. Radiographic evidence of disease progression during or following prior treatment with sorafenib.
12. Patients must have proteinuria < 2+ or a urine protein:creatinine (UPC) ratio < 1.0. Patients who have proteinuria >/= 2+ and UPC ratio >/= 1.0 must undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible.

Exclusion Criteria:

1. Patients who have had prior systemic therapy other than sorafenib. Patients may not have received any systemic chemotherapy </=14 days of Treatment Day 1.
2. Active malignancy other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years.
3. Current, recent (within 4 weeks of Treatment Day 1) or planned participation in an experimental drug study, other than this study.
4. Gastrointestinal disease resulting in an inability to take oral medication or a requirement for intravenous hyperalimentation.
5. History of rupture of existing HCC lesion, or HCC lesion with large necrotic areas seen on conventional imaging studies, as determined by the Principal Investigator, if there is no measurable solid tumor area > 1.5 cm.
6. Inadequately controlled hypertension (defined as systolic blood pressure >140 and/or diastolic blood pressure > 90).
7. Prior history of hypertensive crisis or hypertensive encephalopathy.
8. New York Heart Association Class II or greater congestive heart failure.
9. Cardiac arrhythmia not controlled by medication.
10. History of myocardial infarction or unstable angina within 6 months of Treatment Day 1.
11. History of stroke or transient ischemic attack within 6 months prior to Day 1 of treatment.
12. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1.
13. Evidence of clinically significant [Common Terminology Criteria (CTC) Grade 3 or 4] venous or arterial thrombotic disease within previous 6 months.
14. Radiographic evidence of major tumor thrombus in the vena cava.
15. History of hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1.
16. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
17. History of significant gastrointestinal bleeding requiring procedural intervention (eg variceal banding, Transjugular Intrahepatic Portosystemic Shunts (TIPS) procedure, arterial embolization) within three months prior to treatment day 1. Patients at risk for varices (based on the following: known history of esophageal or gastric varices; evidence of hepatic cirrhosis and/or portal hypertension including biopsy-proven cirrhosis, radiographic evidence of cirrhosis, hypersplenism, or radiographic findings of varices) will be screened for esophageal varices.
18. (Continuation of # 17) If varices are identified that require intervention (banding), that patient will not be eligible for the trial until the varices have been adequately treated.
19. Known CNS disease, except for treated brain metastases. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear accelerator (LINAC), or equivalent) or a combination as deemed appropriate by the treating physician.
20. (Continuation of # 20) Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
21. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study.
22. Core biopsy, fine needle aspiration, or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1.
23. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1.
24. Serious, non-healing wound, active ulcer, or untreated bone fracture.
25. 0ngoing or active infection requiring parenteral therapy.
26. Known HIV disease.
27. Uncontrolled psychiatric illness.
28. Known hypersensitivity to any component of bevacizumab and erlotinib.
29. Pregnancy (positive pregnancy test) or lactation.
30. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kaseb, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kaseb AO, Morris JS, Iwasaki M, Al-Shamsi HO, Raghav KP, Girard L, Cheung S, Nguyen V, Elsayes KM, Xiao L, Abdel-Wahab R, Shalaby AS, Hassan M, Hassabo HM, Wolff RA, Yao JC. Phase II trial of bevacizumab and erlotinib as a second-line therapy for advanced hepatocellular carcinoma. Onco Targets Ther. 2016 Feb 15;9:773-80. doi: 10.2147/OTT.S91977. eCollection 2016. PMID 26929648
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 participants signed consent, 1 patient withdrew consent prior to receiving treatment.
Period: Overall Study
Arm/Group | Erlotinib + Bevacizumab
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib + Bevacizumab
Number analyzed (Participants) | 44
Age, Continuous [Median (Standard Deviation); unit: years] | 63.05 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival is defined as time from initiation of therapy until documented disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 59 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Bevacizumab
Number analyzed (Participants) | 44
months | 43 [28 to 59]

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time between treatment assignment and radiologic progression at 16 weeks as defined by the amendments of the Response Evaluation Criteria in Solid Tumors (RECIST).Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 16 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Bevacizumab
Number analyzed (Participants) | 44
months | 3.9 [2.0 to 8.3]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is the time in months from start of study treatment to date of death due to any cause.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Bevacizumab
Number analyzed (Participants) | 44
months | 9.9 [8.3 to 15.5]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose through 30 days after the last dose of study medication, up to 43 months.
Arm/Group | Erlotinib + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 33/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 40/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Bevacizumab (N=44)
Acneiform Rash (Skin and subcutaneous tissue disorders) | 40
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 24
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Bruising (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 13
Dysphagia (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 4
other (Gastrointestinal disorders) | 6
Lower GI hemorrhage (Gastrointestinal disorders) | 6
Upper GI Hemorrhage (Gastrointestinal disorders) | 1
Fever without neutropenia (General disorders) | 1
Weight Loss (General disorders) | 10
General Disorder, other (General disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Pain (Head) (General disorders) | 7
Pain (Back) (General disorders) | 2
Pain (Abdomen) (General disorders) | 4
Pain (Muscle) (General disorders) | 2
Pain (Other) (General disorders) | 10
Anemia (Investigations) | 3
Elevated transaminase (Investigations) | 5
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 3
Wound Infection (Infections and infestations) | 1
Pul. Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Hyperbilirubinemia (Investigations) | 13
Hypokalemia (Investigations) | 3
Dry Mouth (Gastrointestinal disorders) | 2
Dry Eyes (General disorders) | 1
Hypertension (Vascular disorders) | 7
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypomagnesemia (Investigations) | 7
Nail Changes (Skin and subcutaneous tissue disorders) | 4
Proteinuria (Renal and urinary disorders) | 18
Mucositis (Gastrointestinal disorders) | 25
Taste Changes (Gastrointestinal disorders) | 7
Voice Changes (Nervous system disorders) | 7
Infection (Infections and infestations) | 4
Syncopy attacks (Nervous system disorders) | 1
Thrombus formation (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT01180959/Prot_SAP_000.pdf